CLINICAL TRIAL: NCT03195257
Title: Glucose-Dependent Insulinotropic Polypeptide - Effects on Markers of Bone Turnover in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mikkel Christensen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Christensen, Associate Professor, Principal Investigator, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GIP-T1DM-BTM
Record Dates: First submitted 2017-06-19; First posted 2017-06-22 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Incretins; Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized, double-blinded, cross-over study with 5 study days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hypoglycemia-saline (Placebo Comparator)
  Interventions: Other: Saline
- Hypoglycemia-GIP (Experimental)
  Interventions: Other: GIP
- Hypoglycemia-GLP-1 (Active Comparator)
  Interventions: Other: GLP-1
- Hyperglycemia-GIP (Experimental)
  Interventions: Other: GIP
- Hyperglycemia-Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: GIP — On 3 matched days with 'hypoglycemia' (i.e. plasma glucose clamped between 3-7 mol/L for 120 minutes) either GIP (4 pmol/kg/min), glucagon-like-peptide-1 (GLP-1) (1 pmol/kg/min) or placebo (saline) was administered; and on 2 separately matched days with 'hyperglycemia' (i.e. clamped at 12 mmol/L for 90 minutes) either GIP (4 pmol/kg/min) or saline was administered.
  Other Names: Glucose-Dependent Insulinotropic Polypeptide
  Arms: Hyperglycemia-GIP; Hypoglycemia-GIP
Other: GLP-1 — On 3 matched days with 'hypoglycemia' (i.e. plasma glucose clamped between 3-7 mol/L for 120 minutes) either GIP (4 pmol/kg/min), glucagon-like-peptide-1 (GLP-1) (1 pmol/kg/min) or placebo (saline) was administered; and on 2 separately matched days with 'hyperglycemia' (i.e. clamped at 12 mmol/L for 90 minutes) either GIP (4 pmol/kg/min) or saline was administered.
  Other Names: glucagon-like-peptide-1
  Arms: Hypoglycemia-GLP-1
Other: Saline — On 3 matched days with 'hypoglycemia' (i.e. plasma glucose clamped between 3-7 mol/L for 120 minutes) either GIP (4 pmol/kg/min), glucagon-like-peptide-1 (GLP-1) (1 pmol/kg/min) or placebo (saline) was administered; and on 2 separately matched days with 'hyperglycemia' (i.e. clamped at 12 mmol/L for 90 minutes) either GIP (4 pmol/kg/min) or saline was administered.
  Other Names: placebo
  Arms: Hyperglycemia-Saline; Hypoglycemia-saline

SUMMARY:
Investigate GIP effects on biomarkers involved in bone homeostasis

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes (positive islet cell/ glutamic acid decarboxylase-65 antibodies)
* Patients without measurable beta cell function (i.e. incremental C-peptide below detection limit (<0.16 nmol/l) following an 5 g-iv-arginine stimulation test,

Exclusion Criteria:

* HbA1c >9% (75 mmol/mol),
* standard plasma biochemical measurements outside normal reference interval (alanine aminotransferase, bilirubin, thyroid-stimulating hormone, hemoglobin, creatinine, and spot urine albumin-creatinine ratio);
* an abnormal state of hypoglycemia awareness,
* significant diabetic complications (i.e. proliferative diabetic retinopathy, neuropathy, severe atherosclerosis, heart disease) and,
* treatment with medication (besides insulin) that could not be paused for 12 hours up to and during the days of the experiments.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2012-11-17 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
C-terminal telopeptide of type I collagen (CTX). | 30 minutes intervals, time 0 up to 120 min

SECONDARY OUTCOMES:
Parathyroid hormone (PTH) | 30 minutes intervals, time 0 up to 120 min
N-terminal propeptide of type 1 procollagen (P1NP). | 30 minutes intervals, time 0 up to 120 min

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen MB, Lund A, Calanna S, Jorgensen NR, Holst JJ, Vilsboll T, Knop FK. Glucose-Dependent Insulinotropic Polypeptide (GIP) Inhibits Bone Resorption Independently of Insulin and Glycemia. J Clin Endocrinol Metab. 2018 Jan 1;103(1):288-294. doi: 10.1210/jc.2017-01949. PMID 29099978